CLINICAL TRIAL: NCT04522583
Title: Increased C-reactive Protein Concentrations in Patients Admitted to the Emergency Department With Troponin Level Elevations Aids to Rule Out Coronary Ischemia
Brief Title: Increased CRP Concentrations in Patients Admitted to the Emergency Department With Troponin Elevation Aids to Rule Out Coronary Ischemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-cardiology-1
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Troponin-positive ED patients: All patients admitted to the ED at the Hillel Yaffe Medical Center in Hadera, Israel, in the period 2016-2019 with cTn level higher than the 99th percentile of cTn concentration in the normal population (>0.014 nanogram/milliliter).
  Interventions: Diagnostic Test: Diagnosis of Myocardial Ischemia

INTERVENTIONS:
Diagnostic Test: Diagnosis of Myocardial Ischemia — Discharge diagnosis of myocardial ischemia

SUMMARY:
The investigators hypothesized that the CRP/troponin ratio measured in patients presenting to the ED with elevated troponin levels could differentiate between patients with cardiac ischemia and those who present due to a systemic inflammatory or infectious disease. The aim of the study was to determine the necessary CRP/troponin ratio required to rule out cardiac ischemia in a large ED population and determine its impact on long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ED in the period 2016-2019 with cTn level higher than the 99th percentile of cTn concentration in the normal population (>0.014 nanogram/milliliter).

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ED at the Hillel Yaffe Medical Center, Hadera, during the period 2016-2019 with cTn level higher than the 99th percentile of cTn concentration in the normal population (>0.014 nanogram/milliliter).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the CRP/Troponin ratio | Within 6 months
  The accuracy of the CRP/Troponin ratio in ruling out of myocardial ischemia according to the diagnosis of ischemia/coronary intervention at discharge analyzed by standard statistical measures

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel